CLINICAL TRIAL: NCT03622957
Title: Exploring the Association Between Phthalates Exposure, Measured Through Their Urinary Metabolites, and Renal Function Impairment in Individuals With TYpe 2 Diabetes - Protocol 2
Brief Title: Association Between Phthalates Exposure and Renal Function Impairment in TYpe 2 Diabetes
Acronym: PURITY-2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Pisa (Other)
Collaborators: Istituto di Fisiologia Clinica CNR (Other)
Responsible Party: Principal Investigator, Anna Solini, Associate Professor, MD, PhD, University of Pisa
Other Study IDs: PURITY - Protocol 2
Record Dates: First submitted 2018-08-06; First posted 2018-08-09 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Diabetes Mellitus, Type 2; Albuminuria; Cardiovascular Risk Factor
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Albuminuria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — First morning spot urine sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type 2 diabetes subjects: Type 2 diabetes subjects consecutively referring to Santa Chiara, Pisa diabetes outpatients clinic

SUMMARY:
The global incidence of diabetic nephropathy (DN) is increasing, with no appreciable reduction in the percent of patients progressing toward end stage renal disease (ESRD) and dialysis (Tuttle et al, 2014, Winocour et al, 2018). Therefore, identification of modifiable risk factors and early biomarkers of progressive decline in kidney function is an urgent clinical need. Phthalates are environmental and dietary contaminants with a various array of use that are identified in many consumer and industrial products; among them, di-(2-ethylhexyl) phthalate (DEHP) and its metabolites (mono 2-ethylhexyl phthalate (MEHP), 5OH-MEHP (MEHHP) and 5oxo-MEHP (MEOHP)) are widely used (Kato et al 2004, Braun et al, 2013). They partially distribute to the human tissues and their urinary and serum levels are directly related; therefore, urinary concentration of phthalates is commonly used as proxy of their exposure in humans (Kato et al 2004).

While the association between phthalates exposure and development of T2D is currently being explored (Dong et al 2017, Dales et al, 2018), little is known about their role in DN. Recent observations show that DEHP and its metabolites are associated with a higher prevalence of low-grade albuminuria and in children exposed to higher phthalates concentrations (Trasande et al, 2014, Wu et al, 2018), however such association has yet to be verified in adults. The environmental ubiquity of the phthalates enhances the importance of investigating the potential relation between their exposure and different degrees of renal function. (Kato et al 2004, Kataria et al, 2015).

Given this premise, the investigators will explore this potential association in a population of subjects with T2D consecutively referring to the outpatient diabetes clinic in Santa Chiara Hospital, Pisa, enrolled on a volunteer basis. During their routine visit at Santa Chiara Hospital outpatient diabetes clinic participants will provide the results of blood tests prescribed as per standard clinical practice along with a first morning, overnight fasting, urine sample collected in a phthalates-free container.

The investigators will record the participants' clinical history, physical examination and anthropometric measurements, will measure their renal function, evaluated by eGFR (calculated with the CDK-EPI formula), albumin excretion, fasting glucose, HbA1c%, and the exposure to phthalates, assessed by total concentrations of MEHP, MEOHP, MEHHP and adjusted for urinary creatinine. In this way, the investigators aim to point out the relationship of urinary phthalates with higher degrees of albuminuria and/or lower eGFR after adjustment for all potential confounders, including therapies.

ELIGIBILITY:
Inclusion Criteria:

Age 18-85 years, T2D diagnosis, T2D duration >6 months,

Exclusion Criteria:

occurring acute clinical conditions, eGFR <15 ml/min/1.73m2, BMI > 40 Kg/m2.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetes individuals referring to our outpatient clinics
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-08-10 (Estimated); Primary Completion 2018-09-03 (Estimated); Study Completion 2018-09-03 (Estimated)

PRIMARY OUTCOMES:
Phthalates exposure [ug/g] | Single routine clinical visit
  Concentrations of metabolites of DEHP [ug/ml] in a first morning spot urine sample (obtained during clinical visit) measured by ultra-HPLC coupled with electrospray ionization/quadrupole time-of-flight MS and then normalized for urinary creatinine [g/ml].
Albuminuria [mg/g] | Single routine clinical visit
  Grade of albuminuria measured by albuminuria/creatininuria ratio [mg/g] in a first morning spot urine sample (obtained during clinical visit).
Glomerular Filtration Rate [ml/min/1.73m2] | Single routine clinical visit
  GFR measured by eGFR (calculated with CDK-EPI formula). Creatinine [mg/dL] is measured in a serum sample (obtained during clinical visit). Physiological parameters (age, sex, race) are obtained during clinical visit.

SECONDARY OUTCOMES:
CV Events (Yes/No) | Single routine clinical visit
  History of cardiovascular events (Non fatal: Acute Myocardial infarction, Unstable Angina, Stroke), evaluated by clinical interview during routine clinical visit.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tuttle KR, Bakris GL, Bilous RW, Chiang JL, de Boer IH, Goldstein-Fuchs J, Hirsch IB, Kalantar-Zadeh K, Narva AS, Navaneethan SD, Neumiller JJ, Patel UD, Ratner RE, Whaley-Connell AT, Molitch ME. Diabetic kidney disease: a report from an ADA Consensus Conference. Diabetes Care. 2014 Oct;37(10):2864-83. doi: 10.2337/dc14-1296. PMID 25249672
- [Background] Winocour PH. Diabetes and chronic kidney disease: an increasingly common multi-morbid disease in need of a paradigm shift in care. Diabet Med. 2018 Mar;35(3):300-305. doi: 10.1111/dme.13564. Epub 2018 Jan 8. PMID 29247554
- [Background] Kato K, Silva MJ, Reidy JA, Hurtz D 3rd, Malek NA, Needham LL, Nakazawa H, Barr DB, Calafat AM. Mono(2-ethyl-5-hydroxyhexyl) phthalate and mono-(2-ethyl-5-oxohexyl) phthalate as biomarkers for human exposure assessment to di-(2-ethylhexyl) phthalate. Environ Health Perspect. 2004 Mar;112(3):327-30. doi: 10.1289/ehp.6663. PMID 14998748
- [Background] Braun JM, Sathyanarayana S, Hauser R. Phthalate exposure and children's health. Curr Opin Pediatr. 2013 Apr;25(2):247-54. doi: 10.1097/MOP.0b013e32835e1eb6. PMID 23429708
- [Background] Dong R, Zhao S, Zhang H, Chen J, Zhang M, Wang M, Wu M, Li S, Chen B. Sex Differences in the Association of Urinary Concentrations of Phthalates Metabolites with Self-Reported Diabetes and Cardiovascular Diseases in Shanghai Adults. Int J Environ Res Public Health. 2017 Jun 5;14(6):598. doi: 10.3390/ijerph14060598. PMID 28587233
- [Background] Dales RE, Kauri LM, Cakmak S. The associations between phthalate exposure and insulin resistance, beta-cell function and blood glucose control in a population-based sample. Sci Total Environ. 2018 Jan 15;612:1287-1292. doi: 10.1016/j.scitotenv.2017.09.009. Epub 2017 Sep 8. PMID 28898934
- [Background] Trasande L, Sathyanarayana S, Trachtman H. Dietary phthalates and low-grade albuminuria in US children and adolescents. Clin J Am Soc Nephrol. 2014 Jan;9(1):100-9. doi: 10.2215/CJN.04570413. Epub 2013 Oct 31. PMID 24178978
- [Background] Wu CF, Hsiung CA, Tsai HJ, Tsai YC, Hsieh HM, Chen BH, Wu MT. Interaction of melamine and di-(2-ethylhexyl) phthalate exposure on markers of early renal damage in children: The 2011 Taiwan food scandal. Environ Pollut. 2018 Apr;235:453-461. doi: 10.1016/j.envpol.2017.12.107. Epub 2018 Jan 6. PMID 29310089
- [Background] Kataria A, Trasande L, Trachtman H. The effects of environmental chemicals on renal function. Nat Rev Nephrol. 2015 Oct;11(10):610-25. doi: 10.1038/nrneph.2015.94. Epub 2015 Jun 23. PMID 26100504
- [Derived] Mengozzi A, Carli F, Biancalana E, Della Latta V, Seghieri M, Gastaldelli A, Solini A. Phthalates Exposure as Determinant of Albuminuria in Subjects With Type 2 Diabetes: A Cross-Sectional Study. J Clin Endocrinol Metab. 2019 May 1;104(5):1491-1499. doi: 10.1210/jc.2018-01797. PMID 30462244